CLINICAL TRIAL: NCT05752929
Title: Comparison of 2 Hyperglycemia-correction Scales in Hospitalized Patients in an Institution in Bogotá, Colombia
Brief Title: Comparison of 2 Hyperglycemia-correction Scales in Hospitalized Patients
Acronym: CAPADOCIA1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Clinica San Rafael (Other)
Responsible Party: Principal Investigator, Javier Mauricio Mora Mendez, Principal investigator, cinical professor in internal medicine, Hospital Universitario Clinica San Rafael
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUCSR20161
Record Dates: First submitted 2023-02-07; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Diabete Type 2; Hyperglycemia
Keywords: Diabetes mellitus; hyperglycemia; hospitalization; treatment; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Diabetes Mellitus; Hypoglycemia | interventions — Insulin; Connor-Davidson Resilience Scale

STUDY DESIGN:
Intervention Model Description: Unblinded, randomized, controlled clinical trial in patients with hyperglycemia and type 2 diabetes mellitus hospitalized
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umpierrez (Active Comparator): The Umpierrez sensitive correction scheme correction
  Interventions: Drug: Insulin
- Davidson (Experimental): Davidson correction factor
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: Insulin — correction scheme with Rapid Acting Insulin Analogs according with the Umpierrez sensitive correction scheme
  Other Names: Umpierrez
  Arms: Umpierrez
Drug: insulin — correction scheme with Rapid Acting Insulin Analogs according with the Davidson correction scheme
  Other Names: Davidson
  Arms: Davidson

SUMMARY:
Hyperglycemia in the hospital is associated with multiple adverse outcomes. Previously, the mobile insulin scheme was used for its control. However, in the last decade, several studies have shown that the insulin basal-bolus (basal plus) regimen is associated with better glycemic control and a lower risk of hypoglycemia.

DETAILED DESCRIPTION:
Introduction:

Hyperglycemia in the hospital is associated with multiple adverse outcomes. Previously, the mobile insulin scheme was used for its control. However, in the last decade, several studies have shown that the insulin basal-bolus (basal plus) regimen is associated with better glycemic control and a lower risk of hypoglycemia.

Objective:

To compare the sensitive scheme of Umpierrez and the correction factor suggested by Davidson (1700/total dose of insulin) for the correction of hyperglycemia in patients with type 1 diabetes mellitus.

Methods:

Unblinded, randomized, controlled clinical trial in patients with hyperglycemia and type 2 diabetes mellitus hospitalized at a hospital in Bogotá, Colombia, between 2016 and 2018. A probabilistic sampling with randomly permuted blocks was performed. The Umpierrez sensitive correction scheme and the Davidson correction factor were compared by evaluating glycemic control at 2 and 5 hours, and the presence of hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus who presented hyperglycemia (above 140 mg/dl) located in the general ward, emergency room or hospitalization and who received a basal or basal bolus insulin scheme.

Exclusion Criteria:

* pregnancy, with acute decompensation of diabetes (diabetic ketoacidosis-hyperosmolar state) or type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of paticipants with Glicemic control | 5 hours
  Glycemic control defined as glucose levels between 70 and 180 mg/dl measured with a glucometer

SECONDARY OUTCOMES:
Number of participants with hypoglycemia | 6 hours
  hypoglycemia defined as glucose levels less than 70 mg/dl measured with a glucometer

CONTACTS AND LOCATIONS:
Overall Officials: Javier Mora, Principal Investigator — Hospital Universitario Clinica San Rafael

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Umpierrez GE, Smiley D, Hermayer K, Khan A, Olson DE, Newton C, Jacobs S, Rizzo M, Peng L, Reyes D, Pinzon I, Fereira ME, Hunt V, Gore A, Toyoshima MT, Fonseca VA. Randomized study comparing a Basal-bolus with a basal plus correction insulin regimen for the hospital management of medical and surgical patients with type 2 diabetes: basal plus trial. Diabetes Care. 2013 Aug;36(8):2169-74. doi: 10.2337/dc12-1988. Epub 2013 Feb 22. PMID 23435159
- [Result] Umpierrez GE, Hellman R, Korytkowski MT, Kosiborod M, Maynard GA, Montori VM, Seley JJ, Van den Berghe G; Endocrine Society. Management of hyperglycemia in hospitalized patients in non-critical care setting: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2012 Jan;97(1):16-38. doi: 10.1210/jc.2011-2098. PMID 22223765
- [Result] Davidson PC, Hebblewhite HR, Steed RD, Bode BW. Analysis of guidelines for basal-bolus insulin dosing: basal insulin, correction factor, and carbohydrate-to-insulin ratio. Endocr Pract. 2008 Dec;14(9):1095-101. doi: 10.4158/EP.14.9.1095. PMID 19158048
- [Result] Aschner P, King H, Triana de Torrado M, Rodriguez BM. Glucose intolerance in Colombia. A population-based survey in an urban community. Diabetes Care. 1993 Jan;16(1):90-3. doi: 10.2337/diacare.16.1.90. PMID 8422838
- [Result] Umpierrez GE, Isaacs SD, Bazargan N, You X, Thaler LM, Kitabchi AE. Hyperglycemia: an independent marker of in-hospital mortality in patients with undiagnosed diabetes. J Clin Endocrinol Metab. 2002 Mar;87(3):978-82. doi: 10.1210/jcem.87.3.8341. PMID 11889147
- [Result] Umpierrez GE, Smiley D, Jacobs S, Peng L, Temponi A, Mulligan P, Umpierrez D, Newton C, Olson D, Rizzo M. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes undergoing general surgery (RABBIT 2 surgery). Diabetes Care. 2011 Feb;34(2):256-61. doi: 10.2337/dc10-1407. Epub 2011 Jan 12. PMID 21228246
- [Result] Umpierrez GE, Smiley D, Zisman A, Prieto LM, Palacio A, Ceron M, Puig A, Mejia R. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes (RABBIT 2 trial). Diabetes Care. 2007 Sep;30(9):2181-6. doi: 10.2337/dc07-0295. Epub 2007 May 18. PMID 17513708
- [Result] Escobedo J, Buitron LV, Velasco MF, Ramirez JC, Hernandez R, Macchia A, Pellegrini F, Schargrodsky H, Boissonnet C, Champagne BM; CARMELA Study Investigators. High prevalence of diabetes and impaired fasting glucose in urban Latin America: the CARMELA Study. Diabet Med. 2009 Sep;26(9):864-71. doi: 10.1111/j.1464-5491.2009.02795.x. PMID 19719706